CLINICAL TRIAL: NCT03208712
Title: Pilot Trial of Radium-223 and Atezolizumab in Patients With Urothelial Carcinoma With Bone Metastases Who Have Had Disease Progression After Platinum-Based Chemotherapy
Brief Title: Radium-223 and Atezolizumab in Patients With Urothelial Carcinoma With Bone Metastases Who Have Had Disease Progression After Platinum-Based Chemotherapy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2017.023; HUM00126822 (Other: University of Michigan)
Record Dates: First submitted 2017-07-03; First posted 2017-07-05 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — atezolizumab; Radium-223

STUDY DESIGN:
Intervention Model Description: Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radium-223 and Atezolizumab (Experimental): Radium- 223 IV (55 kBq/kg) every 3 weeks for up to 6 doses
  Atezolizumab 1200 mg IV once every 3 weeks until investigator determined lack of benefit, unacceptable toxicity, or 17 doses
  Interventions: Drug: Atezolizumab; Drug: Radium-223

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab 1200 mg IV once every 3 weeks
Drug: Radium-223 — Radium- 223 IV (55 kBq/kg) every 3 weeks for up to 6 doses

SUMMARY:
This is a single-arm, single-site pilot of Radium-223 (55 kBq/kg) IV q3 weeks for up to 6 doses in combination with Atezolizumab 1200mg IV once every 3 weeks until investigator determined lack of benefit, unacceptable toxicity, or 17 doses in patients with urothelial carcinoma with bone metastases who have disease progression after platinum-containing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histologic diagnosis of urothelial carcinoma with radiologic, histologic or cytologic evidence of metastatic disease.
* Subjects must have at least 1 bone metastasis of any size on imaging.
* ECOG performance status of 0- 2 (Eastern Cooperative Oncology Group Performance Status: an attempt to quantify cancer patients' general well-being and activities of daily life. The score ranges from 0 to 5 where 0 is asymptomatic and 5 is death.)
* Subjects must have progression of disease within 12 months of platinum-containing chemotherapy (chemotherapy could have been given in the neoadjuvant, adjuvant or metastatic settings) for urothelial cancer.
* Adequate organ and marrow function Subjects must have measurable disease on physical exam or imaging per RECIST 1.1 criteria.
* Recovery to baseline or < Grade 1 CTCAE v.4.03 from toxicities related to any prior treatments, unless AE(s) are clinically non-significant and/or stable on supportive therapy
* Patients must be ≥ 2 weeks from most recent systemic therapy or radiation therapy.
* Women of childbearing potential must have a negative serum pregnancy test within 28 days prior to registration.
* Female subjects of childbearing potential and their male partners, and male subjects must be willing to use a highly effective method of contraception from the time consent is signed until 6 months after treatment discontinuation.

Ability to understand and the willingness to sign a written informed consent

* Age ≥ 18 years
* Life expectancy ≥ 12 weeks
* Able to comply with study protocol, in the investigator's judgment

Exclusion Criteria:

* Prior treatment with anti-PD-1/PD-L1, and anti-CTLA-4 is NOT allowed. Prior intravesical BCG therapy is allowed.
* Treatment with any investigational agent or on an interventional clinical trial within 30 days prior to treatment on protocol
* No prior or concurrent malignancy is allowed except for: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, localized or locally advanced prostate cancer definitively treated without recurrence or with biochemical recurrence only, or any other cancer fully treated or from which the subject has been disease-free for at least 2 years.
* Autoimmune diseases such as rheumatoid arthritis or systemic lupus erythematosus. Note: Vitiligo, mild psoriasis (topical therapy only) or hypothyroidism are allowed.
* Need for systemic corticosteroids > 10 mg prednisone daily or equivalent alternative steroid (except physiologic dose for adrenal replacement therapy) or other immunosuppressive agents (such as cyclosporine or methotrexate). Use of topical and inhaled corticosteroids is permitted.
* Any history of allografts
* General Medical Exclusions
* Evidence of significant uncontrolled concomitant disease that could affect compliance with the protocol or interpretation of results, including significant liver disease (such as cirrhosis, uncontrolled major seizure disorder, or superior vena cava syndrome)
* Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to enrollment, unstable arrhythmias, or unstable angina. Patients with known left ventricular ejection fraction (LVEF) <40% will be excluded.
* Severe infection within 4 weeks prior to initiation of study treatment, including but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Treatment with therapeutic oral or IV antibiotics within 14 days prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g. for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 4 weeks prior to initiation of study treatment of anticipation of need for a major surgical procedure during the course of the study other than for diagnosis
* History of severe allergic, anaphylactic or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity or allergy to biopharmaceuticals produced in Chinese hamster ovary cells or any component of the atezolizumab formulation
* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e. bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Positive test for HIV
* Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C.
* Active tuberculosis
* Administration of a live, attenuated vaccine within 4 weeks prior to initiation of study treatment with atezolizumab or anticipation that such a live, attenuated vaccine will be required during the study.
* Bone marrow dysplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2018-08-02 (Actual)

PRIMARY OUTCOMES:
Percent of Patients that respond to Treatment | Up to 52 weeks
  Primary efficacy will be measured by Objective Response Rate (Complete Response + Partial Response). Complete response will be defined as the disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions. Partial Response will be defined as at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. There can be no appearance of new lesions.

SECONDARY OUTCOMES:
Median Overall Survival Time | Up to 52 weeks
Median Progression Free Survival Time | Up to 52 weeks
  Progression-free survival (PFS) is defined as the duration of time from start of treatment to time of progression.
Number of Patients with Complete Response | Up to 52 weeks
  Complete Response (CR): Disappearance of all target lesions, determined by two separate observations conducted not less than 4 weeks apart. There can be no appearance of new lesions.
Change in QOL Score From Baseline | Up to 52 weeks
  Quality of life as assessed by the EORTC QLQ-C30 (A questionnaire developed by the European Organization for Research and Treatment of Cancer to assess the quality of life of cancer patients) at baseline and during treatment will be described using means or medians and associated measures of variability.

CONTACTS AND LOCATIONS:
Overall Officials: Ajjai Alva, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No